CLINICAL TRIAL: NCT00305448
Title: Phase II Study to Evaluate the Efficacy and Tolerability of Fulvestrant 250mg, 250mg (Plus 250mg Loading Regimen) and 500mg in Postmenopausal Women With ER +ve Advanced Breast Cancer Progressing or Relapsing After Previous Endocrine Therapy
Brief Title: A Clinical Trial to Compare Efficacy and Tolerability of Fulvestrant 250mg, 250mg (Plus 250mg Loading Regimen) and 500mg
Acronym: FINDER I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6997C00004; FINDER I
Record Dates: First submitted 2006-03-20; First posted 2006-03-22 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Advanced Breast Cancer; Metastatic Breast Cancer
Keywords: oncology; cancer; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): Fulvestrant 250 mg intramuscular injection
  Interventions: Drug: Fulvestrant
- 2 (Experimental): Fulvestrant 250mg (Plus 250mg Loading Regimen)
  Interventions: Drug: Fulvestrant
- 3 (Experimental): Fulvestrant 500 mg
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — 250 intramuscular injection
  Other Names: Faslodex; ZD9238
  Arms: 1; 2
Drug: Fulvestrant — 500 mg intramuscular injection
  Arms: 3

SUMMARY:
This study will assess the relationship between fulvestrant dose and efficacy, and determine the dosing regimen as a second line therapy for Japanese postmenopausal women with oestrogen receptor positive advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Breast Cancer has continued to grow after having received treatment with an anti-estrogen hormonal treatment such as tamoxifen or an aromatase inhibitor
* Requiring hormonal treatment
* Postmenopausal women defined as a woman who has stopped having menstrual periods

Exclusion Criteria:

* Treatment with more than one previous regimen of systemic anticancer therapy other than endocrine therapy for advanced breast cancer
* Treatment with more than one previous regimen of endocrine therapy for advanced breast cancer
* An existing serious disease, illness, or condition that will prevent participation or compliance with study procedures

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Japan Medical Director, MD, Study Director — AstraZeneca
Locations (35):
- Japan (35):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Asahi, Chiba
  - Research Site, Chiba, Chiba
  - Research Site, Matsuyama, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kitakyushu, Fukuoka
  - Research Site, Kurume, Fukuoka
  - Research Site, Daito, Fukushima
  - Research Site, Kōriyama, Fukushima
  - Research Site, Ōta, Gunma
  - Research Site, Fukuyama, Hiroshima
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Kure, Hiroshima
  - Research Site, Sapporo, Hokkaido
  - Research Site, Amagasaki, Hyōgo
  - Research Site, Matsubaracho, Kagoshima-ken
  - Research Site, Isehara, Kanagawa
  - Research Site, Sagamihara, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Sendai, Miyagi
  - Research Site, Niigata, Niigata
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Kurashiki, Okayama-ken
  - Research Site, Izumisano, Osaka
  - Research Site, Osaka, Osaka
  - Research Site, Sakai, Osaka
  - Research Site, Suita, Osaka
  - Research Site, Morohongō, Saitama
  - Research Site, Shinden, Saitama
  - Research Site, Shizuoka, Shizuoka
  - Research Site, Shimotsuke, Tochigi
  - Research Site, Chūō, Tokyo
  - Research Site, Koto-ku, Tokyo
  - Research Site, Kawasaki

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women with oestrogen receptor positive advanced breast cancer progressing or relapsing after previousendocrine therapy were randomized between 7th March 2006 and 4th September 2007. The trial was conducted in Japan only. One patient randomised to Fulvestrant 500mg was not dosed, so the Safety population has 46 patients for that arm.
Pre-assignment Details: 8 of the 151 enrolled patients were not randomized to treatment groups for the following reasons - 8 patients were incorrectly enrolled (ie did not comply with one or more inclusion / exclusion criteria).
Groups:
- Fulvestrant 250 mg: Fulvestrant 250 mg
- Fulvestrant 250 mg + Loading Dose: Fulvestrant 250 mg + Loading Dose
- Fulvestrant 500 mg: Fulvestrant 500 mg
Period: Overall Study
Arm/Group | Fulvestrant 250 mg | Fulvestrant 250 mg + Loading Dose | Fulvestrant 500 mg
Started | 45 | 51 | 47
Completed | 14 | 17 | 14
Not Completed | 31 | 34 | 33
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Disease Progression | 27 | 31 | 28
Not completed — Subjective Disease Progression | 1 | 2 | 2
Not completed — Tumor Marker Elevation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fulvestrant 250 mg | Fulvestrant 250 mg + Loading Dose | Fulvestrant 500 mg | Total
Number analyzed (Participants) | 45 | 51 | 47 | 143
Age Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (7.4) | 62.4 (9.5) | 62.7 (9.1) | 62.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 51 | 47 | 143
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: An objective response (OR) is defined as a patient having a best overall response of either complete response (CR) or partial response (PR). A patient has best overall response of CR if she had overall response of CR or PR on one visit and met the confirmation criteria per RECIST. ORR is defined as percentage of patients with objective response.
  Each patient with measurable disease at baseline was assessed for OR from the sequence of Response Evaluation Criteria in Solid Tumors (RECIST) scan data up to data cut-off. RECIST scans were performed every 12 weeks (+/- 2weeks) from randomization
Time Frame: baseline and every 12 weeks (+/- 2weeks) from randomization data up to data cut-off (19th march 2008)
Measure: Number; unit: percentage of participants
Arm/Group | Fulvestrant 250 mg | Fulvestrant 250 mg + Loading Dose | Fulvestrant 500 mg
Number analyzed (Participants) | 45 | 51 | 47
percentage of participants | 11.1 | 17.6 | 10.6

2. Secondary Outcome: Time to Progression (TTP)
Description: Time (in days) from randomization until objective disease progression or death (in the absence of objective progression). RECIST tumour assessments carried out every 12 weeks from randomization (+/- 2 weeks) until data cut-off on 19th March 2008.
Time Frame: every 12 weeks from randomization (+/- 2 weeks) until data cut-off (19th march 2008)
Measure: Median (Full Range); unit: days
Arm/Group | Fulvestrant 250 mg | Fulvestrant 250 mg + Loading Dose | Fulvestrant 500 mg
Number analyzed (Participants) | 45 | 51 | 47
days | 169 [30 to 508] | 211 [0 to 426] | 169 [0 to 590]

3. Secondary Outcome: Duration of Response (DoR)
Description: Time from randomisation until objective progression or death (in the absence of objective progression), measured only in those patients who achieved a confirmed Complete Response or confirmed Partial Response.
Time Frame: RECIST tumour assessments carried out every 12 weeks from randomisation (+/- 2 weeks) until data cut-off on19th March 2008.
Reporting Status: Not Posted
Measure: Number; unit: Time (Days) - using Kaplan-Meier method

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: A Clinical Benefit (CB) responder is defined as a patient having a best overall response of Complete response (CR), Partial Response (PR) or Stable disease (SD) provided SD (or better) was present = 154 days from randomization (ie SD = 24 weeks with the 2 week RECIST assessment time window allowed). The Clinical Benefit Rate is the percentage of patients with CB.
Time Frame: every 12 weeks(+/- 2 weeks) from randomization to data up to data cut-off, 19th March 2008.
Measure: Number; unit: percentage of participants
Arm/Group | Fulvestrant 250 mg | Fulvestrant 250 mg + Loading Dose | Fulvestrant 500 mg
Number analyzed (Participants) | 45 | 51 | 47
percentage of participants | 42.2 | 54.9 | 46.8

5. Secondary Outcome: Pharmacokinetic Parameter: Mean Population Clearance, a Measure of the Efficiency With Which Fulvestrant is Eliminated From the Body
Description: The measure of dispersion for mean population clearance is based on the estimated inter-individual variance
Time Frame: Baseline to 12 weeks
Population: Patients who agreed to participate in the PK substudy. The results are based on 148, 122 and 140 plasma-concentration records from patients in the 250 mg, 250 mg + LD and 500 mg treatment arms respectively.
Measure: Mean (Standard Deviation); unit: L/h
Groups:
- Fulvestrant: Fulvestrant
Arm/Group | Fulvestrant
Number analyzed (Participants) | 70
L/h | 34.4 (0.096)

6. Secondary Outcome: Pharmacokinetic Parameter: Mean Volume of Distribution at Steady State, a Measure of the Apparent Volume in the Body Into Which Fulvestrant Distributes
Description: The measure of dispersion for volume of distribution is based on the inter-individual variance estimated for the apparent volume of plasma into which Fulvestrant distributes
Time Frame: Baseline to 12 weeks
Population: Patients who agreed to participate in the PK substudy.
Measure: Mean (Standard Deviation); unit: Vss/F (L)
Arm/Group | Fulvestrant
Number analyzed (Participants) | 70
Vss/F (L) | 35300 (0.175)

ADVERSE EVENTS:
Arm/Group | Fulvestrant 250 mg | Fulvestrant 250 mg + Loading Dose | Fulvestrant 500 mg
Serious Adverse Events (participants affected / at risk) | 2/45 | 5/51 | 1/46
Other Adverse Events (participants affected / at risk) | 44/45 | 49/51 | 44/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant 250 mg (N=45) | Fulvestrant 250 mg + Loading Dose (N=51) | Fulvestrant 500 mg (N=46)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Brain Stem Infarction (Nervous system disorders) | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0
Diverticular Perforation (Gastrointestinal disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Fallopian Tube Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0 | 0
Optic Neuritis (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant 250 mg (N=45) | Fulvestrant 250 mg + Loading Dose (N=51) | Fulvestrant 500 mg (N=46)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 7 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 3
Constipation (Gastrointestinal disorders) | 4 | 7 | 5
Contusion (Injury, poisoning and procedural complications) | 1 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 1
Fatigue (General disorders) | 7 | 7 | 7
Headache (Nervous system disorders) | 3 | 8 | 4
Hot Flush (Vascular disorders) | 8 | 11 | 7
Hypertension (Vascular disorders) | 4 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 3 | 2
Injection Site Erythema (General disorders) | 3 | 2 | 1
Injection Site Induration (General disorders) | 9 | 6 | 10
Injection Site Pain (General disorders) | 14 | 11 | 14
Injection Site Pruritus (General disorders) | 4 | 2 | 4
Insomnia (Psychiatric disorders) | 4 | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 4 | 2 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Nasopharyngitis (Infections and infestations) | 17 | 15 | 16
Nausea (Gastrointestinal disorders) | 11 | 9 | 6
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 4
Pyrexia (General disorders) | 2 | 4 | 5
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 2
Somnolence (Nervous system disorders) | 3 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 3 | 5
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 3 | 3
Weight Decreased (Investigations) | 3 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less